CLINICAL TRIAL: NCT01565330
Title: An Open Label, Parallel Group, Dose Comparison of Safety and Imaging Characteristics of 111 and 370 MBq (3 and 10 mCi) of 18F-AV-45 for Brain Imaging of Amyloid in Healthy Volunteers and Patients With Alzheimer's Disease (AD)
Brief Title: A Study of Two Doses of 18F-AV-45 in Alzheimer's Disease and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A03
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 111 MBq (3 mCi) AD Group (Experimental): Subjects with AD who received 111MBq (3 mCi) of florbetapir F 18; MBq=megabecquerel
  Interventions: Drug: florbetapir F 18
- 111 MBq (3 mCi) Control Group (Experimental): Healthy controls who received 111MBq (3 mCi) of florbetapir F 18
  Interventions: Drug: florbetapir F 18
- 370 MBq (10 mCi) AD Group (Experimental): Subjects with AD who received 370MBq (10 mCi) of florbetapir F 18
  Interventions: Drug: florbetapir F 18
- 370 MBq (10 mCi) Control Group (Experimental): Healthy controls who received 370MBq (10 mCi) of florbetapir F 18.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — single dose IV injection
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study will test two different doses of florbetapir F 18 to determine which dose is best to image amyloid plaques in the brains of Alzheimer's Disease (AD) patients using a positron emission tomography (PET) scanner.

ELIGIBILITY:
Inclusion Criteria (AD group):

* Greater than 50 years of age
* Probable AD according to the National Institute of Neurological and Communication Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* Mild/moderate dementia as evidenced by a Mini-Mental State Examination (MMSE) score ranging from 10 to 24, boundaries included, at screening
* History of cognitive decline gradual in onset and progressive over a period of at least 6 months

Inclusion Criteria (healthy volunteer group):

* 35 to 55 years of age, inclusive
* MMSE of 29 or greater

Exclusion Criteria (both groups):

* Neurodegenerative disorders other than AD, including, but not limited to Parkinson's disease, Pick's disease, fronto-temporal dementia, Huntington's chorea, Down syndrome, Creutzfeldt-Jacob disease, normal pressure hydrocephalus, and progressive supranuclear palsy
* Diagnosis of other dementing / neurodegenerative disease
* Diagnosis of mixed dementia
* Cognitive impairment resulting from trauma, hypoxic damage, vitamin deficiency, brain infection, brain cancer, endocrine disease, or mental retardation
* Clinically significant infarct or possible multi-infarct dementia as defined by the NINCDS criteria
* Evidence on screening MRI or other biomarker that suggests alternate etiology for cognitive deficit (for healthy controls, evidence suggesting the presence of AD pathology)
* Clinically significant psychiatric disease
* History of epilepsy or convulsions
* Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Current clinically significant cardiovascular disease
* Received investigational medication within the last 30 days

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (3):
- United States (3):
  - Research Site, West Palm Beach, Florida
  - Research Site, North East, Maryland
  - Research Site, Clementon, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 111 MBq (3 mCi) AD Group | 111 MBq (3 mCi) Control Group | 370 MBq (10 mCi) AD Group | 370 MBq (10 mCi) Control Group
Started | 5 | 4 | 4 | 7
Completed | 5 | 4 | 4 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 111 MBq (3 mCi) AD Group | 111 MBq (3 mCi) Control Group | 370 MBq (10 mCi) AD Group | 370 MBq (10 mCi) Control Group | Total
Number analyzed (Participants) | 5 | 4 | 4 | 7 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 74.8 (11.01) | 48.0 (6.73) | 76.8 (10.24) | 45.0 (6.88) | 59.4 (17.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 6
  Male | 3 | 3 | 2 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Florbetapir-PET Scan Quality
Description: Visual evaluation of image quality by nuclear medicine specialist blinded to dose and clinical information; reported on a 5-point scale (5=excellent and 1=poor).
Time Frame: 0-90 min after injection
Population: One subject in the 370 MBq (10 mCi) AD Group did not complete all imaging time periods
Measure: Number; unit: florbetapir scans
Groups:
- 111 MBq (3 mCi) AD Group: Subjects with Alzheimer's Disease (AD) who received 111MBq (3 mCi) of florbetapir F 18; MBq=megabecquerel
Arm/Group | 111 MBq (3 mCi) AD Group | 111 MBq (3 mCi) Control Group | 370 MBq (10 mCi) AD Group | 370 MBq (10 mCi) Control Group
Number analyzed (Participants) | 5 | 4 | 4 | 7
florbetapir scans
  1 - Poor | 0 | 0 | 0 | 0
  2 | 1 | 1 | 0 | 0
  3 | 1 | 3 | 2 | 4
  4 | 3 | 0 | 2 | 3
  5 - Excellent | 0 | 0 | 0 | 0

2. Secondary Outcome: Mean Cortical to Cerebellum SUVR
Description: Standardized Uptake Value ratio (SUVR) is the ratio of tracer uptake in predefined cortical regions, relative to uptake in the whole cerebellum.
Time Frame: 0-90 min after injection
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | 111 MBq (3 mCi) AD Group | 111 MBq (3 mCi) Control Group | 370 MBq (10 mCi) AD Group | 370 MBq (10 mCi) Control Group
Number analyzed (Participants) | 5 | 4 | 4 | 7
SUVR | 1.781 (0.217) | 0.968 (0.050) | 1.658 (0.288) | 0.988 (0.093)

ADVERSE EVENTS:
Time Frame: AEs reported within 7 days of injection; SAEs reported within 30 days of injection.
Arm/Group | 111 MBq (3 mCi) AD Group | 111 MBq (3 mCi) Control Group | 370 MBq (10 mCi) AD Group | 370 MBq (10 mCi) Control Group
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 111 MBq (3 mCi) AD Group (N=5) | 111 MBq (3 mCi) Control Group (N=4) | 370 MBq (10 mCi) AD Group (N=4) | 370 MBq (10 mCi) Control Group (N=7)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE IRRITATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days